CLINICAL TRIAL: NCT02059291
Title: A Randomized, Double-blind, Placebo Controlled Study of Canakinumab in Patients With Hereditary Periodic Fevers (TRAPS, HIDS, or crFMF), With Subsequent Randomized Withdrawal/Dosing Frequency Reduction and Open-label Long-term Treatment Epochs
Brief Title: Study of Efficacy and Safety of Canakinumab in Patients With Hereditary Periodic Fevers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885N2301
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Hereditary Periodic Fevers
Keywords: Canakinumab, interleukin-1, Hereditary Periodic Fevers, auto-inflammatory diseases
MeSH Terms: interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- crFMF: 150 mg (Experimental): During Epoch 2, participants received canakinumab 150mg (or 2mg/kg for participants weighing <= 40kg) q4w for 16 weeks. If participants were eligible for blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded uptitration to canakinumab 300 mg q4w from day 29 through day 112. If patients on the highest allowed canakinumab dose of 300 mg (or 4 mg/kg for patients weighing ≤ 40 kg) q4w and re-flared (PGA ≥ 2 and CRP ≥ 30 mg/L) were not eligible for further up-titration.
  Interventions: Drug: Canakinumab
- crCMF: placebo (Placebo Comparator): During epoch 2, participants received matching placebo to canakinumab 150 mg Participants who required blinded escape,they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab.
  150mg, participants were uptitrated to open-label canakinumab 300 mg.
  Interventions: Drug: Placebo
- HIDS/MKD: 150 mg (Experimental): During Epoch 2, participants received canakinumab 150mg (or 2mg/kg for participants weighing <= 40kg) q4w for 16 weeks. If participants were eligible for blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded uptitration to canakinumab 300 mg q4w from day 29 through day 112. If patients on the highest allowed canakinumab dose of 300 mg (or 4 mg/kg for patients weighing ≤ 40 kg) q4w and re-flared (PGA ≥ 2 and CRP ≥ 30 mg/L) were not eligible for further up-titration.
  Interventions: Drug: Canakinumab
- HIDS/MKD: placebo (Placebo Comparator): During epoch 2, participants received matching placebo to canakinumab 150 mg qw4. Participants who required blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28 and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab 150mg, participants were uptitrated to open-label canakinumab 300 mg.
  Interventions: Drug: Placebo
- TRAPS: 150 mg (Experimental): During Epoch 2, participants received canakinumab 150mg (or 2mg/kg for participants weighing <= 40kg) q4w for 16 weeks. If participants were eligible for blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded uptitration to canakinumab 300 mg q4w from day 29 through day 112. If patients on the highest allowed canakinumab dose of 300 mg (or 4 mg/kg for patients weighing ≤ 40 kg) q4w and re-flared (PGA ≥ 2 and CRP ≥ 30 mg/L) were not eligible for further up-titration
  Interventions: Drug: Canakinumab
- TRAPS: placebo (Placebo Comparator): During epoch 2, participants received matching placebo to canakinumab 150 mg qw4. Participants who required blinded escape,they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between Day 8 and 28 and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab 150mg, participants were uptitrated to open-label canakinumab 300 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — Canakinumab solution for subcutaneous injection in vial which contained 150mg/mL canakinumab in 1 mL solution.
  Other Names: ACZ885
  Arms: HIDS/MKD: 150 mg; TRAPS: 150 mg; crFMF: 150 mg
Drug: Placebo — Matching placebo to canakinumab solution for subcutaneous injection
  Arms: HIDS/MKD: placebo; TRAPS: placebo; crCMF: placebo

SUMMARY:
This study is to determine whether canakinumab is able to induce and maintain a clinically meaningful reduction of disease activity in participants with Hereditary Periodic Fevers (HPF) compared to placebo.

DETAILED DESCRIPTION:
This study consists of 3 randomized cohorts (one per condition of colchicine resistant/intolerant Familial Mediterranean Fever (crFMF), Hyper Immunoglobulin D Syndrome (also known as mevalonate kinase deficiency (HIDS/MKD), and Tumor Necrosis Factor Receptor Associated Periodic Syndrome (TRAPS), and 4 study epochs:

1. Epoch 1: a screening epoch to assess participant's eligibility;
2. Epoch 2: a randomized treatment epoch of 16 weeks where participants are randomized to canakinumab 150 mg every 4 weeks (q4w) or to placebo to obtain efficacy and safety data in a double-blind placebo controlled parallel-arm setting. This epoch contained 2 possible escape options :

   1. early blinded escape option for non responders from Day 8 to Day 28 with here an add-on dose of 150mg canakinumab followed by blinded uptitration at the next scheduled visit (Day 29)
   2. late unblinded escape option for non responders from Day 29 to Day 112; with open-label uptitration
3. Epoch 3: a randomized withdrawal epoch of 24 weeks where canakinumab responders from the randomized treatment epoch were re-randomized to canakinumab 150mg q8w or placebo to assess the potential for canakinumab to maintain clinical efficacy at a reduced dosing frequency;
4. Epoch 4: an open-label treatment epoch of 72 weeks to collect long-term

ELIGIBILITY:
Inclusion Criteria: - Patient's written informed consent (or parent's written informed consent in case of pediatric patient) at screening - Male and female patients at least 2 years of age at the time of the screening visit. Male and female patients >28 days but <2 years eligible for open label treatment only. - Confirmed diagnosis and active flare at randomization - CRP >10mg/L at randomization

Exclusion Criteria: - Use of the following therapies (within varying protocol defined timeframes): Corticosteroids, anakinra, canakinumab, rilonacept, tocilizumab, TNF inhibitors, abatacept, tofacitinib, rituximab, leflunomide, thalidomide, cyclosporine, intravenous immunoglobulin, 6-Merceptopurine, azathioprine, cyclophosphamide, or chlorambucil, any other investigational biologics - History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in - situ cervical cancer), treated or untreated - Significant medical diseases, including but not limited to the following: a. History of organ transplantation b. Elevated liver enzymes ≥3x ULN d. Increase in total bilirubin e. Serious hepatic disorder (Child-Pugh scores B or C) f. Chronic Kidney Disease g. Thyroid disease h. Diagnosis of active peptic ulcer disease i. Coagulopathy j. Significant CNS effects including vertigo and dizziness - Any conditions or significant medical problems which immunecompromise the patient and/or places the patient at unacceptable risk for immunomodulatory therapy - Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (57):
- United States (3):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Cleveland, Ohio
- Belgium (5):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
- France (4):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Saint Augustin
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Galway, Ireland
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (10):
  - Novartis Investigative Site, Sciacca, AG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Roma
- Japan (4):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakyo-ku, Kyoto
  - Novartis Investigative Site, Niigata
- Netherlands (2):
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Utrecht
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
- Spain (5):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lausanne, Switzerland
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
- United Kingdom (2):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Gattorno M, Obici L, Penades IC, Kallinich T, Benseler S, Dekker E, Levy J, De Benedetti F, Lachmann H. Long-Term Efficacy and Safety of Canakinumab in Patients With Tumor Necrosis Factor Receptor-Associated Periodic Syndrome: Results From a Phase III Trial. Arthritis Rheumatol. 2024 Feb;76(2):304-312. doi: 10.1002/art.42695. Epub 2023 Dec 8. PMID 37668289
- [Derived] Jeyaratnam J, Simon A, Calvo I, Constantin T, Shcherbina A, Hofer M, Gattorno M, Martini A, Bader-Meunier B, Vastert B, Levy J, Dekker E, de Benedetti F, Frenkel J. Long-term efficacy and safety of canakinumab in patients with mevalonate kinase deficiency: results from the randomised Phase 3 CLUSTER trial. Rheumatology (Oxford). 2022 May 5;61(5):2088-2094. doi: 10.1093/rheumatology/keab696. PMID 34554243
- [Derived] De Benedetti F, Gattorno M, Anton J, Ben-Chetrit E, Frenkel J, Hoffman HM, Kone-Paut I, Lachmann HJ, Ozen S, Simon A, Zeft A, Calvo Penades I, Moutschen M, Quartier P, Kasapcopur O, Shcherbina A, Hofer M, Hashkes PJ, Van der Hilst J, Hara R, Bujan-Rivas S, Constantin T, Gul A, Livneh A, Brogan P, Cattalini M, Obici L, Lheritier K, Speziale A, Junge G. Canakinumab for the Treatment of Autoinflammatory Recurrent Fever Syndromes. N Engl J Med. 2018 May 17;378(20):1908-1919. doi: 10.1056/NEJMoa1706314. PMID 29768139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consists of 4 study epochs. A total of 203 participants ((181randomized + 4 non-randomized open-label participants in Epoch 2) + (18 TRAPS rollover participants from ACZ885D2203 (NCT01242813) and ACZ885D2207M in Epoch 3)) have been enrolled into this study.
Pre-assignment Details: 126 patients, randomized in Epoch 2, were not re-randomized in Epoch 3. These patients were switched to open-label (OL) treatment. Six patients discontinued OL treatment (1 due to physician decision, 1 due to subject/guardian decision, 3 due to lack of efficacy and 1 due to an adverse event).
Groups:
- Epoch 2: crFMF: 150 mg; Epoch 2: HIDS/MKD: 150 mg; Epoch 2: TRAPS: 150 mg: During Epoch 2, participants received canakinumab 150mg (or 2mg/kg for participants weighing <= 40kg) q4w for 16 weeks. If participants were eligible for blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded uptitration to canakinumab 300 mg q4w from day 29 through day 112. If patients on the highest allowed canakinumab dose of 300 mg (or 4 mg/kg for patients weighing ≤ 40 kg) q4w and re-flared (PGA ≥ 2 and CRP ≥ 30 mg/L) were not eligible for further up-titration.
- Epoch 2: crCMF: Placebo: During epoch 2, participants received matching placebo to canakinumab 150 mg Participants who required blinded escape,they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28, and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab.
  150mg, participants were uptitrated to open-label canakinumab 300 mg
- Epoch 2: HIDS/MKD: Placebo: During epoch 2, participants received matching placebo to canakinumab 150 mg qw4. Participants who required blinded escape, they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between day 8 and day 28 and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab 150mg, participants were uptitrated to open-label canakinumab 300 mg.
- Epoch 2: TRAPS: Placebo: During epoch 2, participants received matching placebo to canakinumab 150 mg qw4. Participants who required blinded escape,they received a single add-on dose of canakinumab (150 mg or 2mg/kg for participants weighing <= 40kg) between Day 8 and 28 and then received blinded one dose of placebo and one dose of canakinumab q4w from day 29 through day 112. If flare or re-flare still occurred after receipt of canakinumab 150mg, participants were uptitrated to open-label canakinumab 300 mg.
- Epoch 2: Non-randomized Open Label Treatment - crFMF: Canakinumab-naïve Japanese patients with non-exon 10 mutations received open-label canakinumab 150 mg (or 2 mg/kg for patients weighing
  ≤ 40 kg) q4w .
- Epoch 2: Non-randomized Open Label HIDS/MKD: Participants in the 28 days to less than 2 years old cohort who received open-label canakinumab 150 mg (or 2mg/kg for patients weighing
  ≤ 40 kg) q4w.
- Epoch 2 (Epoch 3) - Non-randomized Open Label TRAPS: Open-label treatment in Epoch 3 was initiated for TRAPS patients who rolled over from CACZ885D2203 or CACZ885D2207M.
- Epoch 3: crFMF Re-randomized From Epoch 2 - 150 mg; Epoch 3: HIDs/MKD Re-randomized From Epoch 2 - 150 mg; Epoch 3: TRAPS Re-randomized From Epoch 2 - 150 mg: Canakinumab responders who were initially randomized to canakinumab 150 mg q4w and did not re-flare in Epoch 2 were re-randomized at the start of Epoch 3 to canakinumab 150 mg q8w for 24 weeks.
- Epoch 3: crFMF Re-randomized From Epoch 2 - Placebo; Epoch 3: HIDS/MKD Re-randomized From Epoch 2 - Placebo; Epoch 3: TRAPS Re-randomized From Epoch 2 - Placebo: Canakinumab responders who were initially randomized to canakinumab 150 mg q4w and did not re-flare in Epoch 2 were re-randomized at the start of Epoch 3 to placebo for 24 weeks.
- Epoch 3: crFMF, HIDS/MKD, TRAPS - Not Re-randomized: All Epoch 2 non-responders were switched to canakinumab q8w at the start of Epoch 3 for 24 weeks,
- Epoch 4: crFMF - Open Label Cumulative Dose <2700 mg; Epoch 4: HIDS/MKD - Open Label Cumulative Dose <2700 mg; Epoch 4: TRAPS - Open Label Cumulative Dose < 2700 mg: During epoch 4, participants received open label treatment according to the dose regimen administered in epoch 3. Cumulative dose received was less than 2700 mg.
- Epoch 4: crFMF - Open Label Cumulative Dose 2700 mg - <5400 mg; Epoch 4: HIDS/MKD - OL Cumulative Dose 2700 - <=5400 mg; Epoch 4: TRAPS - Open Label Cumulative Dose 2700 - <5400 mg: During epoch 4, participants received open label treatment according to the dose regimen administered in epoch 3. Cumulative dose received was >= 2700 mg and < 5400 mg.
- Epoch 4: crFMF - Open Label Cumulative Dose >=5400 mg; Epoch 4: HIDS/MKD - Open Label Cumulative Dose >=5400 mg; Epoch 4: TRAPS - Open Label Cumulative Dose >=5400 mg: During epoch 4, participants received open label treatment according to the dose regimen administered in epoch 3. Cumulative dose received was > 5400 mg.
Period: Epoch 2
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo | Epoch 2: Non-randomized Open Label Treatment - crFMF | Epoch 2: Non-randomized Open Label HIDS/MKD | Epoch 2 (Epoch 3) - Non-randomized Open Label TRAPS | Epoch 3: crFMF Re-randomized From Epoch 2 - 150 mg | Epoch 3: crFMF Re-randomized From Epoch 2 - Placebo | Epoch 3: HIDs/MKD Re-randomized From Epoch 2 - 150 mg | Epoch 3: HIDS/MKD Re-randomized From Epoch 2 - Placebo | Epoch 3: TRAPS Re-randomized From Epoch 2 - 150 mg | Epoch 3: TRAPS Re-randomized From Epoch 2 - Placebo | Epoch 3: crFMF, HIDS/MKD, TRAPS - Not Re-randomized | Epoch 4: crFMF - Open Label Cumulative Dose <2700 mg | Epoch 4: crFMF - Open Label Cumulative Dose 2700 mg - <5400 mg | Epoch 4: crFMF - Open Label Cumulative Dose >=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose <2700 mg | Epoch 4: HIDS/MKD - OL Cumulative Dose 2700 - <=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose >=5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose < 2700 mg | Epoch 4: TRAPS - Open Label Cumulative Dose 2700 - <5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose >=5400 mg
Started | 31 | 32 | 37 | 35 | 22 | 24 | 2 | 2 | 18 (This Epoch 3 group is shown in Epoch 2 to account for the 203 patients enrolled in the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 31 | 31 | 36 | 33 | 22 | 22 | 2 | 1 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Epoch 3
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo | Epoch 2: Non-randomized Open Label Treatment - crFMF | Epoch 2: Non-randomized Open Label HIDS/MKD | Epoch 2 (Epoch 3) - Non-randomized Open Label TRAPS | Epoch 3: crFMF Re-randomized From Epoch 2 - 150 mg | Epoch 3: crFMF Re-randomized From Epoch 2 - Placebo | Epoch 3: HIDs/MKD Re-randomized From Epoch 2 - 150 mg | Epoch 3: HIDS/MKD Re-randomized From Epoch 2 - Placebo | Epoch 3: TRAPS Re-randomized From Epoch 2 - 150 mg | Epoch 3: TRAPS Re-randomized From Epoch 2 - Placebo | Epoch 3: crFMF, HIDS/MKD, TRAPS - Not Re-randomized | Epoch 4: crFMF - Open Label Cumulative Dose <2700 mg | Epoch 4: crFMF - Open Label Cumulative Dose 2700 mg - <5400 mg | Epoch 4: crFMF - Open Label Cumulative Dose >=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose <2700 mg | Epoch 4: HIDS/MKD - OL Cumulative Dose 2700 - <=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose >=5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose < 2700 mg | Epoch 4: TRAPS - Open Label Cumulative Dose 2700 - <5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose >=5400 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 (Presented in Epoch 2.) | 9 | 10 | 6 | 7 | 4 | 5 | 126 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 9 | 10 | 6 | 7 | 3 | 5 | 120 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Epoch 4
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo | Epoch 2: Non-randomized Open Label Treatment - crFMF | Epoch 2: Non-randomized Open Label HIDS/MKD | Epoch 2 (Epoch 3) - Non-randomized Open Label TRAPS | Epoch 3: crFMF Re-randomized From Epoch 2 - 150 mg | Epoch 3: crFMF Re-randomized From Epoch 2 - Placebo | Epoch 3: HIDs/MKD Re-randomized From Epoch 2 - 150 mg | Epoch 3: HIDS/MKD Re-randomized From Epoch 2 - Placebo | Epoch 3: TRAPS Re-randomized From Epoch 2 - 150 mg | Epoch 3: TRAPS Re-randomized From Epoch 2 - Placebo | Epoch 3: crFMF, HIDS/MKD, TRAPS - Not Re-randomized | Epoch 4: crFMF - Open Label Cumulative Dose <2700 mg | Epoch 4: crFMF - Open Label Cumulative Dose 2700 mg - <5400 mg | Epoch 4: crFMF - Open Label Cumulative Dose >=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose <2700 mg | Epoch 4: HIDS/MKD - OL Cumulative Dose 2700 - <=5400 mg | Epoch 4: HIDS/MKD - Open Label Cumulative Dose >=5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose < 2700 mg | Epoch 4: TRAPS - Open Label Cumulative Dose 2700 - <5400 mg | Epoch 4: TRAPS - Open Label Cumulative Dose >=5400 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 43 | 14 | 2 | 18 | 34 | 14 | 31 | 22 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 14 | 2 | 18 | 33 | 14 | 30 | 21 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Epoch 2: Non-randomized Open Label Treatment - crFMF: Canakinumab-naïve Japanese patients with non-exon 10 mutations received open-label canakinumab 150 mg (or 2 mg/kg for patients weighing
  ≤ 40 kg) q4w
- Total: Total of all reporting groups
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo | Epoch 2: Non-randomized Open Label Treatment - crFMF | Epoch 2: Non-randomized Open Label HIDS/MKD | Epoch 2 (Epoch 3) - Non-randomized Open Label TRAPS | Total
Number analyzed (Participants) | 31 | 32 | 37 | 35 | 22 | 24 | 2 | 2 | 18 | 203
Age, Continuous [Median (Full Range); unit: Years]
  crFMF cohort - randomized | 18.0 (15.02) [2 to 60] | 18.0 (13.38) [4 to 69] | NA (NA) [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA (NA) [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA (NA) [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA (NA) [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA [NA to NA] — This row reflects crFMF cohort - randomized data only. | NA [NA to NA] — This row reflects crFMF cohort - randomized data only. | 18 (14.10) [2 to 69]
  HIDS/MKD cohort - randomized | NA (NA) [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | NA (NA) [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | 12.0 (8.49) [2 to 43] | 9.0 (11.64) [3 to 47] | NA (NA) [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | NA (NA) [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | NA [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | NA [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | NA [NA to NA] — This row reflect HIDS/MKD cohort - randomized data only. | 11.0 (10.08) [2 to 47]
  TRAPS cohort - randomized | NA (NA) [NA to NA] — This row reflect TRAPS cohort - randomized data only. | NA (NA) [NA to NA] — This row reflect TRAPS cohort - randomized data only. | NA (NA) [NA to NA] — This row reflect TRAPS cohort - randomized data only. | NA (NA) [NA to NA] — This row reflect TRAPS cohort - randomized data only. | 13.5 (19.22) [3 to 76] | 16.5 (18.25) [2 to 57] | NA [NA to NA] — This row reflect TRAPS cohort - randomized data only. | NA [NA to NA] — This row reflect TRAPS cohort - randomized data only. | NA [NA to NA] — This row reflect TRAPS cohort - randomized data only. | 15.5 (18.55) [2 to 76]
  crFMF - non-randomized | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | 24.5 [20 to 29] | NA [NA to NA] — This row reflects crFMF non-randomized data only. | NA [NA to NA] — This row reflects crFMF non-randomized data only. | 24.5 [20 to 29]
  HIDS/MKD - non-randomized | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | 1.0 [1 to 1] | NA [NA to NA] — This row reflects HIDS/MIK non-randomized data only. | 1.0 [1 to 1]
  roll-over TRAPS - non-randomized | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | NA [NA to NA] — This row reflects roll-over TRAPS non-randomized data only. | 42.5 [15 to 81] | 42.5 [15 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 24 | 19 | 10 | 13 | 2 | 0 | 7 | 104
  Male | 17 | 17 | 13 | 16 | 12 | 11 | 0 | 2 | 11 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2 | 4 | 2 | 1 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 27 | 27 | 34 | 31 | 20 | 18 | 0 | 1 | 16 | 174
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 3 | 3 | 0 | 2 | 0 | 0 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Resolution of Initial Flare and Absence of New Flares up to the End of the Randomized Treatment Epoch (16 Weeks)
Description: Resolution of the initial disease flare is defined as: Physician's Global Assessment of Disease activity (PGA) <2 and C-reactive protein (CRP) within normal range (<= 10 mg/L) or reduction by at least 70% from baseline. The PGA was evaluated by the investigator based on a 5-point scale: 0 = None (no) disease associated with clinical signs and symptoms; 1 = minimal disease associated signs and symptoms; 2 = mild disease associated signs and symptoms; 3 = moderate disease associated signs and symptoms; and 5 = severe disease associated signs and symptoms.
Time Frame: 16 weeks
Population: The Full Analysis Set (FAS), which consisted of all randomized participants in the randomized treatment epoch who received at least one dose of study drug in Epoch 2, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo
Number analyzed (Participants) | 31 | 32 | 37 | 35 | 22 | 24
Percentage of participants | 61.29 | 6.25 | 35.14 | 5.71 | 45.45 | 8.33
Statistical Analysis 1: Comparison: Epoch 2: crFMF: 150 mg vs Epoch 2: crCMF: Placebo; Test type: Superiority; p < 0.0001, Fisher's exact test
Statistical Analysis 2: Comparison: Epoch 2: HIDS/MKD: 150 mg vs Epoch 2: HIDS/MKD: Placebo; Test type: Superiority; p = 0.0020, Fisher's exact test
Statistical Analysis 3: Comparison: Epoch 2: TRAPS: 150 mg vs Epoch 2: TRAPS: Placebo; Test type: Superiority; p = 0.0050, Fisher's exact test

2. Secondary Outcome: Percentage of Participants Who Achieve Physician's Global Assessment (PGA) < 2
Description: The PGA was evaluated by the investigator based on a 5-point scale: 0 = None (no) disease associated with clinical signs and symptoms; 1 = minimal disease associated signs and symptoms; 2 = mild disease associated signs and symptoms; 3 = moderate disease associated signs and symptoms; and 5 = severe disease associated signs and symptoms.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo
Number analyzed (Participants) | 31 | 32 | 37 | 35 | 22 | 24
Percentage of participants | 64.52 | 9.38 | 45.95 | 5.71 | 45.45 | 4.17
Statistical Analysis 1: Comparison: Epoch 2: crFMF: 150 mg vs Epoch 2: crCMF: Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 16.96, 95% CI 2-sided [4.15 to 69.21]
Statistical Analysis 2: Comparison: Epoch 2: HIDS/MKD: 150 mg vs Epoch 2: HIDS/MKD: Placebo; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 13.63, 95% CI 2-sided [2.83 to 65.59]
Statistical Analysis 3: Comparison: Epoch 2: TRAPS: 150 mg vs Epoch 2: TRAPS: Placebo; Test type: Superiority; p = 0.0028, Regression, Logistic; Odds Ratio (OR) = 23.79, 95% CI 2-sided [2.52 to 224.86]

3. Secondary Outcome: Percentage of Participants With the Serologic Remission
Description: Serologic remission was defined as C-reactive protein <= 10 mg/L.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo
Number analyzed (Participants) | 31 | 32 | 37 | 35 | 22 | 24
Percentage of participants | 67.74 | 6.25 | 40.54 | 5.71 | 36.36 | 8.33
Statistical Analysis 1: Comparison: Epoch 2: crFMF: 150 mg vs Epoch 2: crCMF: Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 29.78, 95% CI 2-sided [5.86 to 151.31]
Statistical Analysis 2: Comparison: Epoch 2: HIDS/MKD: 150 mg vs Epoch 2: HIDS/MKD: Placebo; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 12.71, 95% CI 2-sided [2.53 to 63.89]
Statistical Analysis 3: Comparison: Epoch 2: TRAPS: 150 mg vs Epoch 2: TRAPS: Placebo; Test type: Superiority; p = 0.0149, Regression, Logistic; Odds Ratio (OR) = 6.64, 95% CI 2-sided [1.20 to 36.57]

4. Secondary Outcome: Percentage of Participants With Normalized Serum Amyloid A (SAA) Level
Description: Normalized SAA was defined as SAA <= 10 mg/L.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo
Number analyzed (Participants) | 31 | 32 | 37 | 35 | 22 | 24
Percentage of participants | 25.81 | 0.00 | 13.51 | 2.86 | 27.27 | 0.00
Statistical Analysis 1: Comparison: Epoch 2: crFMF: 150 mg vs Epoch 2: crCMF: Placebo; Test type: Superiority; p = 0.0286, Regression, Logistic; Odds Ratio (OR) = 17.46, 95% CI 2-sided [0.92 to 332.92]
Statistical Analysis 2: Comparison: Epoch 2: HIDS/MKD: 150 mg vs Epoch 2: HIDS/MKD: Placebo; Test type: Superiority; p = 0.0778, Regression, Logistic; Odds Ratio (OR) = 5.26, 95% CI 2-sided [0.53 to 51.97]
Statistical Analysis 3: Comparison: Epoch 2: TRAPS: 150 mg vs Epoch 2: TRAPS: Placebo; Test type: Superiority; p = 0.0235, Regression, Logistic; Odds Ratio (OR) = 16.69, 95% CI 2-sided [1.04 to 268.50]

5. Secondary Outcome: Percentage of Participants of Canakinumab Responders From Epoch 2 Who Maintained a Clinically Meaningful Response (Absence of New Flares) (40 Weeks)
Description: A responder was defined as a participant who had no flare between week 16 and week 40.
Time Frame: 40 weeks
Population: The re-randomized set was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoch 2: crFMF: 150 mg | Epoch 2: crCMF: Placebo | Epoch 2: HIDS/MKD: 150 mg | Epoch 2: HIDS/MKD: Placebo | Epoch 2: TRAPS: 150 mg | Epoch 2: TRAPS: Placebo
Number analyzed (Participants) | 9 | 10 | 6 | 7 | 4 | 5
Percentage of participants | 77.8 | 30.0 | 50.0 | 14.3 | 75.0 | 40.0
Statistical Analysis 1: Comparison: Epoch 2: crFMF: 150 mg vs Epoch 2: crCMF: Placebo; Test type: Superiority; p = 0.0513, Regression, Logistic; Odds Ratio (OR) = 8.17, 95% CI 2-sided [0.75 to 113.44]
Statistical Analysis 2: Comparison: Epoch 2: HIDS/MKD: 150 mg vs Epoch 2: HIDS/MKD: Placebo; Test type: Superiority; p = 0.2168, Regression, Logistic; Odds Ratio (OR) = 6.00, 95% CI 2-sided [0.27 to 366.24]
Statistical Analysis 3: Comparison: Epoch 2: TRAPS: 150 mg vs Epoch 2: TRAPS: Placebo; Test type: Superiority; p = 0.3571, Regression, Logistic; Odds Ratio (OR) = 4.50, 95% CI 2-sided [0.15 to 313.49]

ADVERSE EVENTS:
Time Frame: up to week 112
Description: Cohort groups were analyzed according to the occurrence of events corresponding to treatments given during epochs 2, 3 and 4.
  'No medication' events cover events that occurred during epoch 4 when no treatment was given.
Groups:
- Non-randomized Open Label crFMF, HIDS/MKD Patients: Canakinumab-naïve Japanese patients with non-exon 10 mutations with cr-FMF who received open-label canakinumab 150 mg (or 2 mg/kg for patients weighing ≤ 40 kg) q4w; and patients in the 28 days to less than 2 years old cohort with HIDS/MKD who received open-label canakinumab 150 mg (or 2mg/kg for patients weighing
  ≤ 40 kg) q4w
- Non-randomized Open Label TRAPS Patients: Open-label treatment in Epoch 3 was initiated for TRAPS patients who rolled over from CACZ885D2203 or CACZ885D2207M
- Randomized ACZ and Placebo TRAPS Patients - Placebo Events; Randomized ACZ and Placebo TRAPS Patients - ACZ Events; Randomized ACZ and Placebo HIDS/MKD Pts - Placebo Events; Randomized ACZ and Placebo HIDS/MKD Pts - No Medication Events; Randomized ACZ and Placebo HIDS/MKD Patients - ACZ Events; Randomized ACZ and Placebo crFMF Patients - Placebo Events; Randomized ACZ and Placebo crFMF Pts - No Medication Events; Randomized ACZ and Placebo crFMF Patients - ACZ Events: Patients who received ACZ885 and/or placebo during epoch 2 and/or epoch 3.
- Randomized ACZ and Placebo TRAPS Pts - No Medication Events: Patients who received ACZ885 and/or placebo during epoch 2 and/or epoch 3 .
- Any ACZ TRAPS Patients - Placebo Events; Any ACZ TRAPS Patients - no Medication Events; Any ACZ TRAPS Patients - ACZ Events; Any ACZ HIDS/MKD Patients - Placebo Events; Any ACZ HIDS/MKD Patients - No Medication Events; Any ACZ HIDS/MKD Patients - ACZ Events; Any ACZ crFMF Patients - Placebo Events; Any ACZ crFMF Patients - No Medication Events; Any ACZ crFMF Patients - ACZ Events: Patients who received ACZ885 during epoch 2 and/or epoch 3
Arm/Group | Non-randomized Open Label crFMF, HIDS/MKD Patients | Non-randomized Open Label TRAPS Patients | Randomized ACZ and Placebo TRAPS Patients - Placebo Events | Randomized ACZ and Placebo TRAPS Pts - No Medication Events | Randomized ACZ and Placebo TRAPS Patients - ACZ Events | Randomized ACZ and Placebo HIDS/MKD Pts - Placebo Events | Randomized ACZ and Placebo HIDS/MKD Pts - No Medication Events | Randomized ACZ and Placebo HIDS/MKD Patients - ACZ Events | Randomized ACZ and Placebo crFMF Patients - Placebo Events | Randomized ACZ and Placebo crFMF Pts - No Medication Events | Randomized ACZ and Placebo crFMF Patients - ACZ Events | Any ACZ TRAPS Patients - Placebo Events | Any ACZ TRAPS Patients - no Medication Events | Any ACZ TRAPS Patients - ACZ Events | Any ACZ HIDS/MKD Patients - Placebo Events | Any ACZ HIDS/MKD Patients - No Medication Events | Any ACZ HIDS/MKD Patients - ACZ Events | Any ACZ crFMF Patients - Placebo Events | Any ACZ crFMF Patients - No Medication Events | Any ACZ crFMF Patients - ACZ Events
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/18 | 0/46 | 0/46 | 0/46 | 0/72 | 0/72 | 0/72 | 0/63 | 0/63 | 0/63 | 0/61 | 0/61 | 0/61 | 0/71 | 0/71 | 0/71 | 0/61 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/18 | 1/46 | 0/46 | 8/46 | 6/72 | 1/72 | 16/72 | 5/63 | 0/63 | 16/63 | 0/61 | 0/61 | 9/61 | 3/71 | 1/71 | 18/71 | 3/61 | 0/61 | 17/61
Other Adverse Events (participants affected / at risk) | 4/4 | 18/18 | 14/46 | 1/46 | 43/46 | 25/72 | 1/72 | 68/72 | 29/63 | 2/63 | 54/63 | 4/61 | 1/61 | 61/61 | 7/71 | 1/71 | 70/71 | 10/61 | 2/61 | 56/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized Open Label crFMF, HIDS/MKD Patients (N=4) | Non-randomized Open Label TRAPS Patients (N=18) | Randomized ACZ and Placebo TRAPS Patients - Placebo Events (N=46) | Randomized ACZ and Placebo TRAPS Pts - No Medication Events (N=46) | Randomized ACZ and Placebo TRAPS Patients - ACZ Events (N=46) | Randomized ACZ and Placebo HIDS/MKD Pts - Placebo Events (N=72) | Randomized ACZ and Placebo HIDS/MKD Pts - No Medication Events (N=72) | Randomized ACZ and Placebo HIDS/MKD Patients - ACZ Events (N=72) | Randomized ACZ and Placebo crFMF Patients - Placebo Events (N=63) | Randomized ACZ and Placebo crFMF Pts - No Medication Events (N=63) | Randomized ACZ and Placebo crFMF Patients - ACZ Events (N=63) | Any ACZ TRAPS Patients - Placebo Events (N=61) | Any ACZ TRAPS Patients - no Medication Events (N=61) | Any ACZ TRAPS Patients - ACZ Events (N=61) | Any ACZ HIDS/MKD Patients - Placebo Events (N=71) | Any ACZ HIDS/MKD Patients - No Medication Events (N=71) | Any ACZ HIDS/MKD Patients - ACZ Events (N=71) | Any ACZ crFMF Patients - Placebo Events (N=61) | Any ACZ crFMF Patients - No Medication Events (N=61) | Any ACZ crFMF Patients - ACZ Events (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Familial mediterranean fever (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Hyper IgD syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
Tumour necrosis factor receptor-associated periodic syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyserositis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Granulomatous rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized Open Label crFMF, HIDS/MKD Patients (N=4) | Non-randomized Open Label TRAPS Patients (N=18) | Randomized ACZ and Placebo TRAPS Patients - Placebo Events (N=46) | Randomized ACZ and Placebo TRAPS Pts - No Medication Events (N=46) | Randomized ACZ and Placebo TRAPS Patients - ACZ Events (N=46) | Randomized ACZ and Placebo HIDS/MKD Pts - Placebo Events (N=72) | Randomized ACZ and Placebo HIDS/MKD Pts - No Medication Events (N=72) | Randomized ACZ and Placebo HIDS/MKD Patients - ACZ Events (N=72) | Randomized ACZ and Placebo crFMF Patients - Placebo Events (N=63) | Randomized ACZ and Placebo crFMF Pts - No Medication Events (N=63) | Randomized ACZ and Placebo crFMF Patients - ACZ Events (N=63) | Any ACZ TRAPS Patients - Placebo Events (N=61) | Any ACZ TRAPS Patients - no Medication Events (N=61) | Any ACZ TRAPS Patients - ACZ Events (N=61) | Any ACZ HIDS/MKD Patients - Placebo Events (N=71) | Any ACZ HIDS/MKD Patients - No Medication Events (N=71) | Any ACZ HIDS/MKD Patients - ACZ Events (N=71) | Any ACZ crFMF Patients - Placebo Events (N=61) | Any ACZ crFMF Patients - No Medication Events (N=61) | Any ACZ crFMF Patients - ACZ Events (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 18 | 0 | 0 | 5 | 0 | 0 | 4 | 0 | 0 | 18 | 0 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 15 | 2 | 19 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 20
Hyper IgD syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 20 | 0 | 0 | 0
Tumour necrosis factor receptor-associated periodic syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 10 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 10 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye allergy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Scleritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 14 | 3 | 0 | 25 | 4 | 0 | 16 | 1 | 0 | 18 | 1 | 0 | 25 | 1 | 0 | 16
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 5 | 1 | 0 | 14 | 0 | 0 | 6 | 0 | 1 | 6 | 0 | 0 | 14 | 0 | 0 | 6
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 5 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 5 | 0 | 0 | 5
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1 | 1 | 8 | 2 | 0 | 22 | 1 | 0 | 12 | 0 | 1 | 12 | 0 | 0 | 23 | 0 | 0 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 2
Gastric dilatation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 8 | 0 | 0 | 5 | 0 | 0 | 4 | 0 | 0 | 8 | 0 | 0 | 6
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 6 | 2 | 0 | 12 | 1 | 0 | 5 | 0 | 0 | 7 | 1 | 0 | 12 | 0 | 0 | 6
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 6 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 6 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 6 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 6
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 7 | 1 | 0 | 9 | 0 | 0 | 11 | 0 | 0 | 8 | 0 | 0 | 9 | 0 | 0 | 11
Malaise (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 7
Pyrexia (General disorders) | 1 | 5 | 1 | 1 | 14 | 11 | 0 | 39 | 3 | 0 | 13 | 0 | 1 | 19 | 4 | 0 | 40 | 2 | 0 | 13
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 10 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 11 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 3 | 1 | 0 | 2
Cystitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 8 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 0 | 5 | 0 | 1 | 10 | 1 | 0 | 8 | 0 | 0 | 6 | 0 | 1 | 11 | 1 | 0 | 9
Influenza (Infections and infestations) | 1 | 2 | 1 | 0 | 5 | 0 | 0 | 14 | 1 | 0 | 10 | 1 | 0 | 7 | 0 | 0 | 14 | 0 | 0 | 11
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 3
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 3 | 2 | 0 | 3 | 0 | 0 | 5 | 0 | 0 | 3 | 0 | 0 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 9 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 8 | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 8
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 8 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 8 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 0 | 8 | 0 | 0 | 14 | 1 | 0 | 3 | 0 | 0 | 10 | 0 | 0 | 15 | 0 | 0 | 3
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 0 | 8 | 0 | 0 | 4 | 1 | 0 | 3 | 1 | 0 | 8
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 2 | 0 | 10 | 3 | 0 | 22 | 1 | 0 | 12 | 1 | 0 | 13 | 1 | 0 | 22 | 1 | 0 | 12
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 9 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 9
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 7 | 0 | 0 | 6 | 0 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 6
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5 | 1 | 0 | 11 | 0 | 0 | 20 | 0 | 0 | 7 | 1 | 0 | 16 | 0 | 0 | 20 | 0 | 0 | 8
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Serum amyloid A protein increased (Investigations) | 1 | 3 | 2 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 2 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 0 | 6 | 1 | 0 | 18 | 2 | 0 | 11 | 1 | 0 | 11 | 1 | 0 | 18 | 0 | 0 | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 6 | 0 | 0 | 10 | 0 | 0 | 13 | 0 | 0 | 8 | 0 | 0 | 10 | 0 | 0 | 14
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 3 | 0 | 1 | 6 | 1 | 0 | 4 | 0 | 0 | 5 | 0 | 1 | 6 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 7 | 1 | 0 | 7 | 0 | 0 | 7 | 0 | 0 | 7 | 0 | 0 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 5 | 0 | 0 | 7 | 2 | 0 | 8 | 0 | 0 | 8 | 0 | 0 | 7 | 1 | 0 | 9
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4
Headache (Nervous system disorders) | 1 | 2 | 3 | 0 | 12 | 4 | 0 | 30 | 2 | 0 | 16 | 1 | 0 | 14 | 1 | 0 | 31 | 0 | 0 | 16
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 9 | 3 | 0 | 21 | 2 | 0 | 6 | 0 | 0 | 12 | 0 | 0 | 21 | 2 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 6 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 6 | 2 | 0 | 22 | 2 | 0 | 8 | 0 | 0 | 7 | 1 | 0 | 22 | 1 | 0 | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 7 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 7 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 5
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 8 | 1 | 0 | 5 | 1 | 0 | 3 | 0 | 0 | 8 | 0 | 0 | 5 | 0 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 3 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT02059291/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02059291/SAP_001.pdf